CLINICAL TRIAL: NCT00896428
Title: Effects of Gallopamil on Bronchial Smooth Muscle Remodelling in Severe Asthma: a Double Blind Study.
Brief Title: Effects of Gallopamil in Severe Asthma
Acronym: REMODEL'ASTHME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX2008/09
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: Asthma; gallopamil; airway remodelling; smooth muscle
MeSH Terms: conditions — Asthma; Airway Remodeling | interventions — Gallopamil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 16 patients with a diagnosis of severe asthma under gallopamil treatment
  Interventions: Drug: Methoxyverapamil (gallopamil)
- 2 (Placebo Comparator): 16 patients with a diagnosis of severe asthma under placebo treatment
  Interventions: Drug: Placebo.

INTERVENTIONS:
Drug: Methoxyverapamil (gallopamil) — 200 mg/day (1 tablet 100 mg morning and evening) for 12 months.
  Arms: 1
Drug: Placebo. — 1 tablet morning and evening for 12 months
  Arms: 2

SUMMARY:
Severe asthma is a difficult to treat disease, characterized by bronchial remodelling, which is an abnormal repair process that contributes to the development of poorly reversible airway narrowing. Such remodelling is now considered as one of the main prognostic factors. Gallopamil-sensitive calcium influx plays a key role in this remodelling process in vitro. The objective of this study is to compare the effects of gallopamil versus placebo on the bronchial smooth muscle remodelling in severe asthmatic patients.

DETAILED DESCRIPTION:
Bronchial remodelling mainly involves an increased mass of bronchial smooth muscle (BSM), which is related with an increase proliferation of smooth muscle cells. Recently, using BSM cells obtained from severe asthmatics, we have demonstrated that such an increase proliferation was induced by an activation cascade (Trian, J Exp Med, 2007). It first started with a gallopamil-sensitive calcium influx which induced the activation of calcium-calmodulin kinase IV (CamK-IV). CamK-IV then enhanced mitochondrial biogenesis through the subsequent activation of various transcription factors including PGC-1α, NRF-1 and mt-TFA. BSM cell proliferation was mainly mitochondria-dependent in vitro in severe asthma whereas that of controls was virtually mitochondria-independent. However, in vivo effects of gallopamil remain to be investigated. We will thus enrol 32 severe asthmatic patients in a phase 2 randomized double blind study against placebo and evaluate the effect of gallopamil on BSM remodelling. Since inflammation also activates mitochondrial biogenesis in BSM cells, we will initially optimized asthma treatment for 3 months by both controlling co morbidities and decreasing bronchial inflammation using exhaled NO and eosinophil count within the induced sputum. We will then perform fiberoptic fibroscopy before and after 12 month treatment with gallopamil.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 18 years
* Written informed consent
* Diagnosis of severe asthma according to ATS criteria

Exclusion Criteria:

* Smoker or former smoker
* Chronic viral infections (hepatitis, HIV)
* Aspergillosis
* Pregnancy
* Breastfeeding
* Contraindications to gallopamil or bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Bronchial smooth muscle remodelling assessed by optic microscopy. | Before and after 12 months treatment.

SECONDARY OUTCOMES:
Bronchial smooth muscle remodelling assessed by electron microscopy | Before and after 12 months treatment.
Bronchial smooth muscle mitochondrial number and activity assessed in vitro | Before and after 12 months treatment.
Bronchial thickness assessed by 3D analysis of computed tomography | Before and after 12 months treatment.
Asthma control using asthma control questionnaire, inflammation monitoring, number of hospitalizations, number of emergency visits, number of unplanned medical visits. | Once per month for 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Berger, Professor, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Hôpital Haut-Lévêque - Centre Hospitalier Universitaire de Bordeaux, Pessac, France

REFERENCES:
- [Background] Trian T, Benard G, Begueret H, Rossignol R, Girodet PO, Ghosh D, Ousova O, Vernejoux JM, Marthan R, Tunon-de-Lara JM, Berger P. Bronchial smooth muscle remodeling involves calcium-dependent enhanced mitochondrial biogenesis in asthma. J Exp Med. 2007 Dec 24;204(13):3173-81. doi: 10.1084/jem.20070956. Epub 2007 Dec 3. PMID 18056286
- [Derived] Girodet PO, Dournes G, Thumerel M, Begueret H, Dos Santos P, Ozier A, Dupin I, Trian T, Montaudon M, Laurent F, Marthan R, Berger P. Calcium channel blocker reduces airway remodeling in severe asthma. A proof-of-concept study. Am J Respir Crit Care Med. 2015 Apr 15;191(8):876-83. doi: 10.1164/rccm.201410-1874OC. PMID 25633090